CLINICAL TRIAL: NCT07337109
Title: A Longitudinal Study Evaluating Oral-Health-Related Quality of Life and Treatment Patterns Among Dentin Hypersensitivity Sufferers in the Real World
Brief Title: A Study Evaluating Oral-Health-Related Quality of Life and Treatment Patterns Among Dentin Hypersensitivity Sufferers
Status: Recruiting | Type: Observational
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Other Study IDs: 400318
Record Dates: First submitted 2025-12-12; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- New sufferers of self-reported Dentin Hypersensitivity aged 18+ years

SUMMARY:
The primary purpose of this study is to characterize changes in Oral-Health-Related Quality of Life (OHrQoL), as measured by the Dentin Hypersensitivity Experience Questionnaire (DHEQ) over a 12-month period.

DETAILED DESCRIPTION:
This will be a longitudinal study investigating OHrQoL and treatment patterns amongst new sufferers of self-reported Dentin Hypersensitivity (DH). Over the 12-month study duration, 375 participants suffering from DH will complete questionnaires online once per month.

ELIGIBILITY:
Inclusion Criteria:

* Participant who has provided consent indicating they have been informed of all pertinent aspects of the study.
* All genders who, at the time of screening, are aged more than or equal to (>=)18 years.
* Anyone who has begun to experience dentin hypersensitivity (self-reported) within the past three months.
* Anyone who has started to use products to treat their tooth sensitivity within the past three months.
* Participant who is able to independently complete all activities online.
* Participants residing in the United States.

Exclusion Criteria:

* Anyone who has any chronic health conditions that could impact their participation in this study, such as cancer, mental health disorders, history of serious illness in the last three months, history of substance abuse, or planned surgery during the study period.
* Participant whose sensitivity could be caused by other factors or clinical pathology than DH, as self-reported on the screening questionnaire, which include:

  1. Anyone who suffers from tooth cavities, significant gum disease, cracked or fractured teeth, temporomandibular joint disease (TMD), or who has had tooth extractions or fillings within the last three months.
  2. Anyone who wears braces (including Invisalign-like appliances) for treatment or dentures (full or partial).
  3. Participant who has undergone treatment for periodontal or gum disease within 6 months of screening or is currently undergoing treatment for periodontal or gum disease.
  4. Participant who has been informed by a Dental Health Care Professional (DHCP) that they have active periodontitis.
  5. Participant who has been informed by a DHCP that they have active caries.
  6. Participant with any chronic and/or severe painful health condition(s) which lead to regular use of pain relief medications (more than 3 days a week).
* Anyone who has participated in another dentin hypersensitivity study within the last three months.
* Currently participating in another research study or will be participating in any other research study at any point during this study's duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who are new sufferers of DH and have begun treating their DH.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Total DHEQ Score Over 12 Months | Baseline and up to 12 Months
  Change from baseline in total DHEQ score and each of the domain scores (daily restrictions, coping behaviors, personal identity, social impact, emotional impact) over 12 months. The DHEQ has total 15 questions each will be scored on a scale ranging from 1 (strongly disagree) to 7 (strongly agree), thus total possible score will be ranging from 15 to 105, where higher score indicates worst outcome.

SECONDARY OUTCOMES:
Description of Treatment Selection Over 12 Months | Up to 12 Months
  Participants will select the appropriate options from the given list of products. Data will be summarized using descriptive statistics.
Treatment Discontinuation/Switch Over 12 Months | Up to 12 Months
  Participant will respond to the question either as Yes or No. Data will be summarized using descriptive statistics.
Frequency of Treatment Used Over 12 Months | Up to 12 Months
  Participants will select the appropriate frequency options from the given list. Data will be summarized using descriptive statistics.
Frequency of DH Over 12 Months | Up to 12 Months
  Participants will select the appropriate frequency options from the given list. Data will be summarized using descriptive statistics.
Frequency of Brushing at Baseline, Months 6 and 12 | Baseline, Months 6 and 12
  Participants will select the appropriate frequency options from the given list. Data will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs (Virtual Site), Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No